CLINICAL TRIAL: NCT01338740
Title: Prospective Study to Assess the Efficacy of Switching to Infliximab in Moderately to Severely Active Chrohn's Disease Patients With Primary Non-response or Loss of Response to Adalimumab
Brief Title: Switching From Adalimumab to Infliximab
Acronym: ADA-IFX
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: 2010/566
Record Dates: First submitted 2011-04-18; First posted 2011-04-19 (Estimated); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Crohn's Disease
Keywords: Chrohn's disease; Moderate to severely active Crohn's disease patients
MeSH Terms: conditions — Crohn Disease | interventions — Adalimumab; Infliximab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — At regular intervals, the results of interim blood tests will be documented (3x).
  After 10, 26 and 52 weeks, additional serum samples will be taken for determination of antibodies against Adalimumab and Infliximab. The serum levels of Adalimumab (week 0) and Infliximab (week 10, 26 and 52) will be determined.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Switch from Adalimumab to Infliximab: Moderately to severely active Crohn's disease patients with primary non-response or loss of response to Adalimumab, will switch to Infliximab.
  Interventions: Drug: Adalimumab and Infliximab

INTERVENTIONS:
Drug: Adalimumab and Infliximab — Patients with moderately to severely active Crohn's disease with primary non-response or loss of response to Adalimumab switch to Infliximab.

SUMMARY:
Switching to Adalimumab has proven to be efficacious in Crohn's disease (CD) patients with intolerance or loss of response to Infliximab. Currently there are no studies on the efficacy of switching to Infliximab in patients with loss of response or primary non-response to Adalimumab. Even in rheumatology, where switching between all classes of anti-TNFα biologicals is common practice, there are no scientific data on switching from humanized to chimeric anti-TNFα antibodies.

The purpose of this study is to document the efficacy of such a switch and to identify the possible predictive factors for success.

If treatment with Adalimumab fails (despite optimal dose and interval) and the treating physician therefore decided to switch to infliximab, the patient may be enrolled in this observational study. At regular intervals (every Remicade), the patient will be clinically re-evaluated. The disease activity score will be calculated: Crohn's disease activity index (CDAI). At regular intervals, the results of interim blood tests will be documented (3x). The succession will be 1 year. At week 10, 26 and 52, additional serum samples will be taken for determination of antibodies against Adalimumab and Infliximab. The serum levels of Adalimumab (week 0) and Infliximab (week 10, 26 and 52) will be determined.

For this study there is no specific therapy change. The study wants only to document the results of a therapy switch that, in current clinical practice, is made by the treating physician.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Crohn's disease confirmed by radiological, endoscopical or histological evidence.
* Moderately to severely active Crohn's disease: Crohn's Disease Activity Index (CDAI) ≥ 220 ≤ 450, scored during the screening period.
* Primary non-response to Adalimumab induction (160mg at week 0, 80 mg at week 2, then 40 mg every 2 weeks: q2w), defined as CDAI ≥ 220 in combination with C-Reactive Protein (CRP) ≥ 0.5mg/dl or endoscopic or radiological evidence of disease activity and evaluated 2 weeks after 6 injections (q2w) of Adalimumab (injections week 0 to week 10, evaluation week 12). OR Loss of response to Adalimumab, defined as CDAI ≥ 220 in combination with CRP ≥ 0.5mg/dl or endoscopic or radiological evidence of disease activity and after at least 4 weeks of weekly injections of Adalimumab (40mg).
* Male or female aged 18-75 years old.
* No history, signs or symptoms of active or latent, untreated tuberculosis (TB).
* Having laboratory results as follows:

Serum Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) levels not exceeding 2 times the upper limit of normal for the central laboratory conducting the test Serum creatinine not exceeding 1.7 mg/dl. Platelets ≥ 100 x 103 cells/µl. Neutrophils ≥ 1.5 x 103 cells/µl.

* Having met all concomitant medication criteria:

Capable of providing informed consent, prior to any study related procedure.

Exclusion Criteria:

* Exclusively fistulising Crohn's disease or exclusive involvement of the upper gastrointestinal (GI) tract.
* Subject with abscess or suspicion of abscess.
* Subject with obstructive fibrotic strictures (with prestenotic dilatation).
* Subject with short bowel syndrome.
* Subject who has had a surgical bowel resection within the past 6 months or planning of any resection at the time while enrolled in the study.
* Subject with Ulcerative Colitis or Indeterminant Colitis.
* Subject with ostomy or ileoanal pouch.
* Subject who is currently receiving total parenteral nutrition.
* Subject who has previously been treated with Infliximab or Certolizumab Pegol.
* Subject with positive stool cultures for enteric pathogens or positive C. difficile toxins during screening period.
* Subject who has received any investigational drug within 12 weeks prior to screening.
* Subject with a history of drug or alcohol abuse within the past 3 years.
* Females who are pregnant or breast feeding.
* Females of child bearing age not practicing effective birth control.
* Subject with a history of malignancy irrespective of time (except carcinoma- in situ of cervix or basal cell carcinoma or squamous cell carcinoma that was successfully treated).
* Subject with a history or symptoms of lymphoproliferative disease.
* Subject with a history of Human Immunodeficiency Virus (HIV), chronic or active Hepatitis B.
* History of Congestive Heart Failure (CHF), including medically controlled asymptomatic CHF.
* Subject who currently has or had an opportunistic infection (e.g. cytomegalovirus (CMV), pneumocystis carinii, aspergillosis, histoplasmosis, coccidioidomycosis) within 6 months prior to screening.
* Subject who currently has an active infection.
* Subject who has a transplanted organ (except for corneal transplant).
* History of known demyelinating disease such as optic neuritis or multiple sclerosis.
* Signs or symptoms of severe, progressive or uncontrolled renal, hepatic, hematologic, gastrointestinal, endocrine, pulmonary, cardiac, neurologic, psychiatric or cerebral disease.

CONCOMITANT MEDICATION

1. Corticosteroids (prednisone, (methyl)prednisolone, budesonide):

   stable dose for 2 weeks prior to baseline, then tapering at the discretion of the investigator.
2. Immunosuppressants (azathioprine, 6-mercaptopurine, methotrexate):

   patients taking this medication prior to baseline: stable dose for 8 weeks prior to baseline, then stable dose until week 26 of the study. Starting or restarting of immunosuppressants is allowed until week 2, then stable dose until week 26 of the study.
3. 5-ASA analogues (sulphasalazine, mesalazine): stable dose for 4 weeks prior to baseline, stable dose until week 26 of the study.
4. Antibiotics (e.g. quinolone, metronidazole): stable dose for 2 weeks prior to baseline.
5. Adalimumab: at least 2 week washout period prior to first Infliximab infusion.

Starting or increasing the dose of other medication for Crohn's disease than Infliximab during the study will be considered as "treatment failure". (except for immunosuppressants as described above under 2.)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with moderately to severely active Crohn's disease with primary non-response or loss of response to Adalimumab, switch to Infliximab.
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2014-02-17 (Actual); Study Completion 2014-02-17 (Actual)

PRIMARY OUTCOMES:
Assess efficacy of switching from Adalimumab to Infliximab. | after 10 weeks
  The primary objective of the study is to assess the efficacy of switching to Infliximab for the induction of clinical remission in subjects with moderately to severely active Crohn's disease with primary non-response or loss of response to Adalimumab.
  The proportion of subjects achieving clinical remission at week 10 after 3 infusions of Infliximab (week 0, 2 and 6). Clinical remission is defined as a total Crohn's Disease Activity Index (CDAI) score of 150 or less.

SECONDARY OUTCOMES:
induction of clinical response | after 10 weeks
  To assess the efficacy of switching from Adalimumab to Infliximab for the induction of clinical response. The proportion of subjects with clinical response (at least 70 point decrease in Crohn's Disease Activity Index (CDAI)) at week 10.
induction of strong clinical response | after 10 weeks
  To assess the efficacy of switching from Adalimumab to Infliximab for the induction of strong clinical response.
  The proportion of subjects with strong clinical response (at least 100 point decrease in CDAI) at week 10.
Sustained Clinical Response | after 26 and 52 weeks
  To assess the efficacy of switching from Adalimumab to Infliximab to achieve sustained clinical response, treating with maintenance Infliximab infusions.
  The proportion of subjects with sustained clinical response (at least 100 and 70 point decrease in CDAI) at weeks 26 and 52.
Sustained Clinical Remission | after 26 and 52 weeks
  To assess the efficacy of switching from Adalimumab to Infliximab to achieve sustained clinical remission, treating with maintenance Infliximab infusions.
  The proportion of subjects with sustained clinical remission (CDAI 150 or less) at weeks 26 and 52.
Induction and maintenance of steroid-free remission. | after 10, 26 and 52 weeks
  To assess the efficacy of switching from Adalimumab to Infliximab for the induction and maintenance of steroid-free remission.
  The proportion of subjects with steroid-free remission (CDAI 150 or less) at weeks 10, 26 and 52.
Sustained clinical remission without need for Infliximab therapy optimization. | after 26 and 52 weeks
  To assess the efficacy of switching from Adalimumab to Infliximab to achieve sustained clinical remission, treating with maintenance Infliximab infusions, without the need for Infliximab therapy optimization (interval shortening or dose increase).
  The proportion of subjects with sustained clinical remission (CDAI 150 or less) at weeks 26 and 52, without the need for Infliximab therapy optimization (interval shortening or dose increase).
Treatment failure | during 52 weeks
  To assess the treatment failure of switching from Adalimumab to Infliximab. The proportion of patients with treatment failure. Failure is defined as cessation of Infliximab due to intolerance or insufficient efficacy despite therapy optimization or the start or dose increase of any other Crohn's disease medication during the study (including corticosteroids, immunosuppressants and 5-aminosalicylic acid (5-ASA) analogues).
Tolerance and safety for switching from Adalimumab to Infliximab. | After 10, 26 and 52 weeks.
  Adverse events/Serious adverse events will be analysed. Hematology and biochemistry will be analysed at weeks 10, 26 and 52.
Serological factors associated with switching from Adalimumab to Infliximab. | after 10, 26 and 52 weeks
  * C-Reactive Protein (CRP) at screening, weeks 10, 26 and 52.
  * Antibodies to Adalimumab at baseline, weeks 10, 26 and 52.
  * Trough level of Adalimumab at baseline.
  * Antibodies to Infliximab at weeks 10, 26 and 52.
  * Trough level of Infliximab at weeks 10, 26 and 52.

CONTACTS AND LOCATIONS:
Overall Officials: Harald Peeters, Ph.D., M.D., Principal Investigator — University Hospital, Ghent
Locations (16):
- Belgium (16):
  - Sint-Augustinus, Antwerp
  - UZ Antwerpen, Antwerp
  - Imelda Hospital, Bonheiden
  - Cliniques Universitaires Saint-Luc, Brussels
  - ULB université libre (erasme), Brussels
  - Ziekenhuis Oost-Limburg, Genk
  - University Hospital Ghent, Ghent
  - Virga Jesse hospital, Hasselt
  - AZ Groeninge, Kortrijk
  - UZ Leuven, Leuven
  - CHC (Centre Hospitalier Chrétien), Liège
  - CHU de liège, Liège
  - Hospital Maas en kempen, Maaseik
  - AZ Damiaan, Ostend
  - Clinique Saint-Pierre, Ottignies
  - Heilig Hartziekenhuis Roeselare, Roeselare

REFERENCES:
- See also: Related Info — http://www.uzgent.be